CLINICAL TRIAL: NCT01788163
Title: A Diagnostic Study to Determine the Prevalence of EGFR Mutations in Asian and Russian Patients With Advanced NSCLC of Adenocarcinoma and Non-adenocarcinoma Histologies
Brief Title: Asia Pacific and Russia Diagnostic Study for EGFR Testing
Acronym: IGNITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D7913C00074
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: EGFR Mutation Status in aNSCLC Patients
Keywords: EGFR; aNSCLC; mutation status; diagnostic study; Russia; China; Asia
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Locally advanced/metastatic NSCLC pats. (Other): Patients with locally advanced (stage IIIA/B) or metastatic NSCLC who have not received any local or systemic chemotherapy, and are not eligible for curative treatment (including surgery and chemoradiotherapy)
  Interventions: Genetic: EGFR mutation test

INTERVENTIONS:
Genetic: EGFR mutation test — EGFR mutation being tested in tissue and blood
  Other Names: Determination of EGFR mutation done at the Pathology lab

SUMMARY:
Interventional diagnostic, international, multicenter and non-comparative study of EGFR mutation status in aNSCLC patients (locally advanced and/or metastatic disease) with adenocarcinoma and non-adenocarcinoma histologies. It will be conducted in Asia Pacific and Russia and will assess the current status of EGFR mutation testing, and the concordance of EGFR mutation status derived from tumour samples and blood based circulating free DNA.

DETAILED DESCRIPTION:
A diagnostic study to determine the prevalence of EGFR mutations in Asian and Russian patients with advanced NSCLC of Adenocarcinoma and Non-adenocarcinoma histologies

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed locally advanced NSCLC (stage IIIA/B) not suitable for curative treatment or metastatic (stage IV) NSCLC
* Newly diagnosed patients with locally advanced and/or metastatic NSCLC who are systemic treatment Naive (i.e. no chemotherapy or EGFR-TKI) or patients with recurrent disease who have previously received adjuvant chemotherapy (not including EGFR-TKI)
* Provision of diagnostic cancer tissue or cytology sample upon inclusion (surgical specimen, biopsy sample, or cytology sample is acceptable) and Provision of a routine blood (plasma) sample in China, Russia, Taiwan and Korea
* Patients aged 18 years and older

Exclusion Criteria:

* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease)
* Evidence of any other significant clinical disorder or laboratory finding that made it undesirable for the patient to participate in the study
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Actual)
Dates: Start 2013-02-27 (Actual); Primary Completion 2014-08-25 (Actual); Study Completion 2016-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rose McCormack, PhD, Study Director — AstraZeneca, PHB
Locations (71):
- Australia (9):
  - Research Site, Campbelltown, New South Wales
  - Research Site, Coffs Harbour, New South Wales
  - Research Site, Concord, New South Wales
  - Research Site, Tamworth, New South Wales
  - Research Site, Tweed Heads, New South Wales
  - Research Site, Wahroonga, New South Wales
  - Research Site, Brisbane, Queensland
  - Research Site, Woolloongabba, Queensland
  - Research Site, Murdoch, Western Australia
- China (14):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Changzhou
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Foshan
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Suzhou
  - Research Site, Taiyuan
  - Research Site, Wuhan
  - Research Site, Zhengzhou
- Indonesia (2):
  - Research Site, Jakarta
  - Research Site, Surabaya
- Research Site, Kuala Lumpur, Malaysia
- Russia (35):
  - Research Site, Arkhangelsk
  - Research Site, Barnaul
  - Research Site, Belgorod
  - Research Site, Birobidzhan
  - Research Site, Chelyabinsk
  - Research Site, Chita
  - Research Site, Irkutsk
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Khabarovsk
  - Research Site, Khanty-Mansiysk
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Lipetsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Oryol
  - Research Site, Perm
  - Research Site, Pyatigorsk
  - Research Site, Rostov-on-Don
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Surgut
  - Research Site, Tula
  - Research Site, Ufa
  - Research Site, Veliky Novgorod
  - Research Site, Vladivostok
  - Research Site, Volgograd
  - Research Site, Yakutsk
  - Research Site, Yaroslavl
  - Research Site, Yuzhno-Sakhalinsk
- Research Site, Singapore, Singapore
- South Korea (3):
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Seoul
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Tainan
  - Research Site, Taipei
- Thailand (3):
  - Research Site, Chiang Mai
  - Research Site, Khon Kaen
  - Research Site, Patumwan Bangkok

REFERENCES:
- See also: D7913C00074_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=599&filename=D7913C00074Ignite%20Extension%20Obversational%20CSR_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Males or females that had Stage IIIB or Stage IV adenocarcinoma of the lung and who were systemic treatment naive or patients with recurrent disease who have previously received adjuvant chemotherapy were enrolled 27 February 2013 and 25 July 2014. The study was carried out in Asiapac countries and Russia.
Pre-assignment Details: A total of 3500 patients were initially enrolled, of which 118 patients were enrolled but were excluded from the study upon failure to satisfy all eligibility criteria. These patients were not included in any analysis data sets.
Groups:
- China: Subjects in China that meet Inclusion/Exclusion (I/E) and population criteria.
- Taiwan: Subjects in Taiwan that meet I/E and population criteria
- South Korea: Subjects in South Korea that meet I/E and population criteria
- Australia: Subjects in Australia that meet I/E and population criteria
- Thailand: Subjects in Thailand that meet I/E and population criteria
- Singapore: Subjects in Singapore that meet I/E and population criteria
- Malaysia: Subjects in Malaysia that meet I/E and population criteria
- Indonesia: Subjects in Indonesia that meet I/E and population criteria
- Russia: Subjects in Russia that meet I/E and population criteria
Period: Overall Study
Arm/Group | China | Taiwan | South Korea | Australia | Thailand | Singapore | Malaysia | Indonesia | Russia
Started | 1458 | 271 | 62 | 71 | 94 | 102 | 50 | 302 | 972
Completed | 1403 | 271 | 62 | 71 | 94 | 95 | 49 | 254 | 956
Not Completed | 55 | 0 | 0 | 0 | 0 | 7 | 1 | 48 | 16
Not completed — Other | 53 | 0 | 0 | 0 | 0 | 7 | 1 | 48 | 15
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- China: Subjects in China that meet I/E and population criteria.
- Total: Total of all reporting groups
Arm/Group | China | Taiwan | South Korea | Australia | Thailand | Singapore | Malaysia | Indonesia | Russia | Total
Number analyzed (Participants) | 1458 | 271 | 62 | 71 | 94 | 102 | 50 | 302 | 972 | 3382
Age, Continuous [Mean (Standard Deviation); unit: Years] — Calculated from birth date to screening visit date
  Years
    Age (years) | 59.8 (10.57) | 66.4 (12.66) | 65.9 (11.91) | 67.1 (10.02) | 61.2 (12.3) | 63.3 (10.79) | 58.7 (10.5) | 57.1 (11.46) | 59.8 (8.9) | 60.4 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants] — Frequency distribution of Male/Female
  Participants
    Female | 535 | 111 | 22 | 36 | 40 | 42 | 14 | 97 | 245 | 1142
    Male | 923 | 160 | 40 | 35 | 54 | 60 | 36 | 205 | 727 | 2240

OUTCOME MEASURES:

1. Primary Outcome: Overall Tumour Epidermal Growth Factor Receptor (EGFR) Mutation Status
Description: The 95% Confidence intervals were calculated using Clopper Pearson method for each country.
Time Frame: At Screening
Population: Tumour Evaluable Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | China | Taiwan | South Korea | Australia | Thailand | Singapore | Malaysia | Indonesia | Russia
Number analyzed (Participants) | 1391 | 271 | 62 | 58 | 87 | 100 | 49 | 273 | 924
Percentage of participants
  Mutation Negative | 59.2 [56.6 to 61.8] | 52.0 [45.9 to 58.1] | 77.4 [65.0 to 87.1] | 70.7 [57.3 to 81.9] | 71.3 [60.6 to 80.5] | 45.0 [35.0 to 55.3] | 65.3 [50.4 to 78.3] | 57.5 [51.4 to 63.4] | 88.1 [85.8 to 90.1]
  Mutation Positive | 40.8 [38.2 to 43.4] | 48.0 [41.9 to 54.1] | 22.6 [12.9 to 35.0] | 29.3 [18.1 to 42.7] | 28.7 [19.5 to 39.4] | 55.0 [44.7 to 65.0] | 34.7 [21.7 to 49.6] | 42.5 [36.6 to 48.6] | 11.9 [9.9 to 14.2]

2. Primary Outcome: Tumour EGFR Mutation by Subtype
Description: Frequency distribution of subjects with a positive mutation status by the mutation subtype and country.
Time Frame: At Screening
Population: Tumour Evaluable Population
Measure: Number; unit: Participants
Arm/Group | China | Taiwan | South Korea | Australia | Thailand | Singapore | Malaysia | Indonesia | Russia
Number analyzed (Participants) | 1391 | 271 | 62 | 58 | 87 | 100 | 49 | 273 | 924
Participants
  G719x mutation only | 8 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Exon 19 deletion only | 283 | 61 | 5 | 12 | 13 | 27 | 7 | 43 | 63
  Exon 19 deletion +T790M | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Exon 19 deletion + other | 6 | 1 | 0 | 0 | 0 | 5 | 0 | 0 | 8
  Exon 19 Other only | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  T790M only | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  T790M + other | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Exon 20 insertions only | 11 | 2 | 1 | 0 | 2 | 3 | 2 | 0 | 0
  L858R mutation only | 239 | 57 | 7 | 4 | 7 | 17 | 8 | 70 | 26
  S768I mutation only | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  L858R mutation + other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  L861Q mutation only | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 3 | 2
  Exon 21 Other only | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 6
  Other | 6 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 2

3. Primary Outcome: Tumour EGFR Mutation Status by Histology
Description: Only subjects who had a recorded Histological Type of Adenocarcinoma or Non-adenocarcinoma are included. Confidence intervals were calculated using Clopper Pearson method for each country.
Time Frame: At Screening
Population: Tumour Evaluable Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- China-Adenocarcinoma: Subjects in China that meet I/E and population criteria with a histological type of Adenocarcinoma.
- China-Non-adenocarcinoma: Subjects in China that meet I/E and population criteria with a histological type of Non-Adenocarcinoma.
- Taiwan-Adenocarcinoma: Subjects in Taiwan that meet I/E and population criteria with a histological type of Adenocarcinoma.
- Taiwan-Non-adenocarcinoma: Subjects in Taiwan that meet I/E and population criteria with a histological type of Non-Adenocarcinoma.
- South Korea-Adenocarcinoma: Subjects in South Korea that meet I/E and population criteria with a histological type of Adenocarcinoma.
- South Korea-Non-adenocarcinoma: Subjects in South Korea that meet I/E and population criteria with a histological type of Non-Adenocarcinoma.
- Australia-Adenocarcinoma: Subjects in Australia that meet I/E and population criteria with a histological type of Adenocarcinoma.
- Australia-Non-adenocarcinoma: Subjects in Australia that meet I/E and population criteria with a histological type of Non-Adenocarcinoma.
- Thailand-Adenocarcinoma: Subjects in Thailand that meet I/E and population criteria with a histological type of Adenocarcinoma.
- Thailand-Non-adenocarcinoma: Subjects in Thailand that meet I/E and population criteria with a histological type of Non-Adenocarcinoma.
- Singapore-Adenocarcinoma: Subjects in Singapore that meet I/E and population criteria with a histological type of Adenocarcinoma.
- Singapore-Non-adenocarcinoma: Subjects in Singapore that meet I/E and population criteria with a histological type of Non-Adenocarcinoma.
- Malaysia-Adenocarcinoma: Subjects in Malaysia that meet I/E and population criteria with a histological type of Adenocarcinoma.
- Malaysia-Non-adenocarcinoma: Subjects in Malaysia that meet I/E and population criteria with a histological type of Non-Adenocarcinoma.
- Indonesia-Adenocarcinoma: Subjects in Indonesia that meet I/E and population criteria with a histological type of Adenocarcinoma.
- Indonesia-Non-adenocarcinoma: Subjects in Indonesia that meet I/E and population criteria with a histological type of Non-Adenocarcinoma.
- Russia-Adenocarcinoma: Subjects in Russia that meet I/E and population criteria with a histological type of Adenocarcinoma.
- Russia-Non-adenocarcinoma: Subjects in Russia that meet I/E and population criteria with a histological type of Non-Adenocarcinoma.
Arm/Group | China-Adenocarcinoma | China-Non-adenocarcinoma | Taiwan-Adenocarcinoma | Taiwan-Non-adenocarcinoma | South Korea-Adenocarcinoma | South Korea-Non-adenocarcinoma | Australia-Adenocarcinoma | Australia-Non-adenocarcinoma | Thailand-Adenocarcinoma | Thailand-Non-adenocarcinoma | Singapore-Adenocarcinoma | Singapore-Non-adenocarcinoma | Malaysia-Adenocarcinoma | Malaysia-Non-adenocarcinoma | Indonesia-Adenocarcinoma | Indonesia-Non-adenocarcinoma | Russia-Adenocarcinoma | Russia-Non-adenocarcinoma
Number analyzed (Participants) | 1026 | 361 | 208 | 61 | 46 | 15 | 49 | 7 | 73 | 13 | 95 | 3 | 40 | 6 | 212 | 59 | 500 | 402
Percentage of participants
  Mutation Negative | 48.7 [45.6 to 51.8] | 88.9 [85.2 to 92.0] | 42.8 [36.0 to 49.8] | 83.6 [71.9 to 91.8] | 69.6 [54.2 to 82.3] | 100.0 [78.2 to 100.0] | 67.3 [52.5 to 80.1] | 85.7 [42.1 to 99.6] | 69.9 [58.0 to 80.1] | 84.6 [54.6 to 98.1] | 43.2 [33.0 to 53.7] | 66.7 [9.4 to 99.2] | 62.5 [45.8 to 77.3] | 83.3 [35.9 to 99.6] | 54.7 [47.8 to 61.5] | 67.8 [54.4 to 79.4] | 82.0 [78.3 to 85.3] | 96.3 [93.9 to 97.9]
  Mutation Positive | 51.3 [48.2 to 54.4] | 11.1 [8.0 to 14.8] | 57.2 [50.2 to 64.0] | 16.4 [8.2 to 28.1] | 30.4 [17.7 to 45.8] | 0.0 [0.0 to 21.8] | 32.7 [19.9 to 47.5] | 14.3 [0.4 to 57.9] | 30.1 [19.9 to 42.0] | 15.4 [1.9 to 45.4] | 56.8 [46.3 to 67.0] | 33.3 [0.8 to 90.6] | 37.5 [22.7 to 54.2] | 16.7 [0.4 to 64.1] | 45.3 [38.5 to 52.2] | 32.2 [20.6 to 45.6] | 18.0 [14.7 to 21.7] | 3.7 [2.1 to 6.1]

4. Primary Outcome: Overall Plasma EGFR Mutation Status
Description: Plasma samples were only performed in China, Taiwan, South Korea and Russia. The Confidence intervals were calculated using Clopper Pearson method for each country.
Time Frame: At Screening
Population: Plasma Evaluable Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | China | Taiwan | South Korea | Russia
Number analyzed (Participants) | 1421 | 271 | 61 | 941
Percentage of participants
  Mutation Negative | 79.3 [77.1 to 81.4] | 73.1 [67.4 to 78.3] | 86.9 [75.8 to 94.2] | 90.8 [88.7 to 92.5]
  Mutation Positive | 20.7 [18.6 to 22.9] | 26.9 [21.7 to 32.6] | 13.1 [5.8 to 24.2] | 9.2 [7.5 to 11.3]

5. Primary Outcome: Plasma EGFR Mutation by Subtype
Description: Plasma samples were only performed in China, Taiwan, South Korea and Russia. Frequency distribution of subjects with a positive mutation status by the mutation subtype and country.
Time Frame: At Screening
Population: Plasma Evaluable Population
Measure: Number; unit: Participants
Arm/Group | China | Taiwan | South Korea | Russia
Number analyzed (Participants) | 1421 | 271 | 61 | 941
Participants
  G719X mutation only | 5 | 0 | 0 | 0
  Exon 19 deletion only | 152 | 35 | 1 | 61
  Exon 19 deletion + other | 0 | 1 | 0 | 0
  T790M + other | 2 | 0 | 0 | 0
  Exon 20 insertions only | 4 | 2 | 0 | 1
  L858R mutation only | 122 | 30 | 6 | 25
  S768I mutation only | 2 | 1 | 0 | 0
  L858R mutation + Other | 0 | 1 | 0 | 0
  L861Q mutation only | 4 | 1 | 0 | 0
  Other | 3 | 2 | 1 | 0

6. Primary Outcome: Plasma EGFR Mutation Status by Histology
Description: as for outcome 3
Time Frame: At Screening
Population: Plasma Evaluable Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | China-Adenocarcinoma | China-Non-Adenocarcinoma | Taiwan-Adenocarcinoma | Taiwan-Non-adenocarcinoma | South Korea-Adenocarcinoma | South Korea-Non-adenocarcinoma | Russia-Adenocarcinoma | Russia-Non-adenocarcinoma
Number analyzed (Participants) | 1047 | 369 | 208 | 61 | 46 | 15 | 513 | 409
Percentage of participants
  Mutation Negative | 74.4 [71.6 to 77.0] | 93.2 [90.2 to 95.6] | 68.3 [61.5 to 74.5] | 90.2 [79.8 to 96.3] | 82.6 [68.6 to 92.2] | 100.0 [78.2 to 100.0] | 89.3 [86.3 to 91.8] | 92.9 [90.0 to 95.2]
  Mutation Positive | 25.6 [23.0 to 28.4] | 6.8 [4.4 to 9.8] | 31.7 [25.5 to 38.5] | 9.8 [3.7 to 20.2] | 17.4 [7.8 to 31.4] | 0.0 [0.0 to 21.8] | 10.7 [8.2 to 13.7] | 7.1 [4.8 to 10.0]

7. Secondary Outcome: Concordance Rate of Comparison of Mutation Status Between Tumour and Plasma Samples
Description: Plasma samples were only performed in China, Taiwan, South Korea and Russia.
Time Frame: At Screening
Population: Tumour and Plasma Evaluable Population
Measure: Number; unit: Percentage
Arm/Group | China | Taiwan | South Korea | Russia
Number analyzed (Participants) | 1355 | 271 | 61 | 894
Percentage | 77.6 [75.2 to 79.8] | 76.8 [71.3 to 81.6] | 83.6 [71.9 to 91.8] | 85.8 [83.3 to 88.0]

8. Secondary Outcome: Sensitivity and Specificity of Comparison of Mutation Status Between Tumour and Plasma Samples
Description: Plasma samples were only performed in China, Taiwan, South Korea, and Russia. Participants only include those who had sensitivity and specificity tests performed.
Time Frame: At Screening
Population: Tumour and Plasma Evaluable Population
Measure: Number; unit: Percentage
Groups:
- China - Sensitivity: Subjects in China that meet I/E and population criteria, who had a sensitivity test performed.
- China - Specificty: Subjects in China that meet I/E and population criteria, who had a specificity test performed.
- Taiwan - Sensitivity: Subjects in Taiwan that meet I/E and population criteria, who had a sensitivity test performed.
- Taiwan - Specificity: Subjects in Taiwan that meet I/E and population criteria, who had a specificity test performed.
- South Korea - Sensitivity: Subjects in South Korea that meet I/E and population criteria, who had a sensitivity test performed.
- South Korea - Specificity: Subjects in South Korea that meet I/E and population criteria, who had a specificity test performed.
- Russia - Sensitivity: Subjects in Russia that meet I/E and population criteria, who had a sensitivity test performed.
- Russia - Specificity: Subjects in Russia that meet I/E and population criteria, who had a specificity test performed.
Arm/Group | China - Sensitivity | China - Specificty | Taiwan - Sensitivity | Taiwan - Specificity | South Korea - Sensitivity | South Korea - Specificity | Russia - Sensitivity | Russia - Specificity
Number analyzed (Participants) | 548 | 807 | 130 | 141 | 14 | 47 | 109 | 785
Percentage | 48.7 | 97.1 | 53.8 | 97.9 | 42.9 | 95.7 | 30.3 | 93.5

9. Secondary Outcome: Predictive Values of Comparison of Mutation Status Between Tumour and Plasma Samples
Description: Plasma samples were only performed in China, Taiwan, South Korea, and Russia. Participants include only those who had Positive and Negative Predictive tests performed.
Time Frame: At Screening
Population: Tumour and Plasma Evaluable Population
Measure: Number; unit: Percentage
Groups:
- China - Positive Predictive Value: Subjects in China that meet I/E and population criteria, who had a Positive Predictive test performed.
- China - Negative Predictive Value: Subjects in China that meet I/E and population criteria, who had a Negative Predictive test performed.
- Taiwan - Positive Predictive Value: Subjects in Taiwan that meet I/E and population criteria, who had a Positive Predictive test performed.
- Taiwan - Negative Predictive Value: Subjects in Taiwan that meet I/E and population criteria, who had a Negative Predictive test performed.
- South Korea - Positive Predictive Value: Subjects in South Korea that meet I/E and population criteria, who had a Positive Predictive test performed.
- South Korea - Negative Predictive Value: Subjects in South Korea that meet I/E and population criteria, who had a Negative Predictive test performed.
- Russia - Positive Predictive Value: Subjects in Russia that meet I/E and population criteria, who had a Positive Predictive test performed.
- Russia - Negative Predictive Value: Subjects in Russia that meet I/E and population criteria, who had a Negative Predictive test performed.
Arm/Group | China - Positive Predictive Value | China - Negative Predictive Value | Taiwan - Positive Predictive Value | Taiwan - Negative Predictive Value | South Korea - Positive Predictive Value | South Korea - Negative Predictive Value | Russia - Positive Predictive Value | Russia - Negative Predictive Value
Number analyzed (Participants) | 290 | 1065 | 73 | 198 | 8 | 53 | 84 | 810
Percentage | 92.1 | 73.6 | 95.9 | 69.7 | 75.0 | 84.9 | 39.3 | 90.6

10. Secondary Outcome: Tumour EGFR Mutation Testing
Description: Frequencies of tumour EGFR mutation testing practices parameters.
Time Frame: At Screening
Population: Enrolled Population
Measure: Number; unit: Participants
Arm/Group | China | Taiwan | South Korea | Australia | Thailand | Singapore | Malaysia | Indonesia | Russia
Number analyzed (Participants) | 1458 | 271 | 62 | 71 | 94 | 102 | 50 | 302 | 972
Participants
  Tumour Sample | 1394 | 271 | 62 | 60 | 92 | 101 | 49 | 273 | 936
  Mutation Test Not Performed | 64 | 0 | 0 | 11 | 2 | 1 | 1 | 29 | 36

11. Secondary Outcome: Tumour EGFR Mutation Testing Rates
Description: Testing Success rate is the percentage of subjects with a non-missing test result. Mutation Detection Rate is the percentage of subjects with successful test that detects a mutation.
Time Frame: At Screening
Population: Enrolled Population
Measure: Number; unit: Percentage of Participants
Arm/Group | China | Taiwan | South Korea | Australia | Thailand | Singapore | Malaysia | Indonesia | Russia
Number analyzed (Participants) | 1458 | 271 | 62 | 71 | 94 | 102 | 50 | 302 | 972
Percentage of Participants
  Testing Success Rate | 99.8 | 100.0 | 100.0 | 96.7 | 94.6 | 99.0 | 100.0 | 100.0 | 98.7
  Mutation Detection Rate | 40.7 | 48.0 | 24.2 | 28.3 | 27.2 | 54.5 | 34.7 | 42.5 | 12.7

12. Secondary Outcome: Tumour EGFR Mutation Testing Turnaround Time
Description: Tumour EGFR mutation testing turnaround time is the number of days from the test request to getting the test result.
Time Frame: At Screening
Population: Enrolled Population
Measure: Mean (Standard Deviation); unit: Time (Days)
Arm/Group | China | Taiwan | South Korea | Australia | Thailand | Singapore | Malaysia | Indonesia | Russia
Number analyzed (Participants) | 1458 | 271 | 62 | 71 | 94 | 102 | 50 | 302 | 972
Time (Days) | 6.2 (5.34) | 7.4 (12.29) | 11.7 (12.70) | 12.9 (8.19) | 70.8 (43.85) | 8.4 (4.90) | 8.6 (3.55) | 6.5 (2.33) | 14.3 (26.84)

13. Secondary Outcome: Plasma EGFR Mutation Testing
Description: Plasma samples were only performed in China, Taiwan, South Korea and Russia. Frequencies of plasma EGFR mutation testing practices parameters.
Time Frame: At Screening
Population: Enrolled Population
Measure: Number; unit: Participants
Arm/Group | China | Taiwan | South Korea | Russia
Number analyzed (Participants) | 1458 | 271 | 62 | 972
Participants
  Plasma Sample | 1421 | 271 | 62 | 950
  Mutation Test Not performed | 37 | 0 | 0 | 22

14. Secondary Outcome: Plasma EGFR Mutation Testing Rates
Description: Testing Success rate is the percentage of subjects with a non-missing test result. Mutation Detection Rate is the percentage of subjects with successful test that detects a mutation. Plasma samples were only performed in China, Taiwan, South Korea and Russia.
Time Frame: At Screening
Population: Enrolled Population
Measure: Number; unit: Percentage of Participants
Arm/Group | China | Taiwan | South Korea | Russia
Number analyzed (Participants) | 1458 | 271 | 62 | 972
Percentage of Participants
  Testing Success Rate | 100.0 | 100.0 | 98.4 | 99.1
  Mutation Detection Rate | 20.7 | 26.9 | 12.9 | 9.2

15. Secondary Outcome: Plasma EGFR Mutation Testing Turnaround Time
Description: Plasma samples were only performed in China, Taiwan, South Korea and Russia. Plasma EGFR mutation testing turnaround time is the number of days from the test request to getting the test result.
Time Frame: At Screening
Population: Enrolled Population
Measure: Mean (Standard Deviation); unit: Time (Days)
Arm/Group | China | Taiwan | South Korea | Russia
Number analyzed (Participants) | 1458 | 271 | 62 | 972
Time (Days) | 39.8 (44.24) | 26.7 (12.62) | 18.1 (13.72) | 90.1 (105.69)

16. Secondary Outcome: Demographics and Disease Characteristics by Tumour EGFR Mutation Status
Description: Correlation of demographic and disease characteristics are summarized by EGFR mutation status with results from a multivariate logistic regression using stepwise forward selection with a 10% significance level for model entry.
Time Frame: At Screening
Population: Tumour Evaluable Population
Measure: Number; unit: Participants
Groups:
- EGFR Mutation Positive: Participants who were EGFR Mutation Positive for the analysis population.
- EGFR Mutation Negative: Participants who were EGFR Mutation Negative for the analysis population.
Arm/Group | EGFR Mutation Positive | EGFR Mutation Negative
Number analyzed (Participants) | 1051 | 2164
Participants
  Histology: Adenocarcinoma | 952 | 1297
  Histology: Non-adenocarcinoma | 89 | 838
  Smoking Status: Never-Smoker | 705 | 647
  Smoking Status: Ever-Smoker | 346 | 1517
  Gender: Male | 480 | 1647
  Gender: Female | 571 | 517
  Region: Asia Pacific | 941 | 1350
  Region: Russia | 110 | 814
  Age: <=65 | 695 | 1447
  >65 | 356 | 717
  World Health Organization Performance Status: 0-1 | 866 | 1808
  World Health Organization Performance Status: 2 | 128 | 276
  Current Disease Status: IIIA | 42 | 266
  Current Disease Status: IIIB | 86 | 371
  Current Disease Status: IV | 923 | 1527
  Number of Organs with Metastasis = 1 | 458 | 901
  Number of Organs with Metastasis = 2 | 266 | 408
  Number of Organs with Metastasis = 3 | 127 | 149
  Number of Organs with Metastasis = 4 | 53 | 61
  Number of Organs with Metastasis = 5 | 16 | 15
  Number of Organs with Metastasis = 6 | 2 | 2
  Number of Organs with Metastasis = 7 | 3 | 1
Statistical Analysis 1: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0001, Regression stepwise — Histology: Adenocarcinoma vs Non-adenocarcinoma; 10% significance level for entry criteria; Wald Chi Square Statistic = 81.1237
Statistical Analysis 2: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0001, Regression stepwise — Histology: Adenocarcinoma vs Non-adenocarcinoma; 10% significance level for model entry; Odds Ratio (OR) = 3.973
Statistical Analysis 3: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0075, Regression Stepwise — Gender: Male vs. Female; 10% significance level for entry criteria; Wald Chi Square Statistic = 7.1526
Statistical Analysis 4: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0075, Regression Stepwise — Gender: Male vs. Female; 10% Significance Level for model entry; Odds Ratio (OR) = 1.409
Statistical Analysis 5: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0001, Regression Stepwise — Smoking Status: Never-smoker vs. Ever-smoker; 10% significance level for entry criteria; Wald Chi Square Statistic = 51.8456
Statistical Analysis 6: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0001, Regression Stepwise — Smoking Status: Never-smoker vs. Ever-smoker; 10% Significance Level for model entry; Odds Ratio (OR) = 2.515
Statistical Analysis 7: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0001, Regression Stepwise — Region: Asia Pacific vs. Russia; 10% Significance Level for entry criteria; Wald Chi Square Statistic = 98.1065
Statistical Analysis 8: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0001, Regression Stepwise — Region: Asia Pacific vs. Russia; 10% Significance Level for model entry; Odds Ratio (OR) = 3.929
Statistical Analysis 9: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0909, Regression Stepwise — Number of organs with metastasis; 10% significance level for entry criteria; Wald Chi Square Statistic = 2.8589
Statistical Analysis 10: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0909, Regression Stepwise — Number of organs with metastasis; 10% significance level for model entry; Odds Ratio (OR) = 1.086

17. Secondary Outcome: Time Since First Non-small-cell Lung Carcinoma (NSCLC) Diagnosis by Tumor EGFR Mutation
Description: Number of months since the first diagnosis of NSCLC from informed consent date.
Time Frame: At Screening
Population: Tumour Evaluable Population
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | EGFR Mutation Positive | EGFR Mutation Negative
Number analyzed (Participants) | 1051 | 2164
Months | 2.6 (8.93) | 2.6 (9.79)

18. Secondary Outcome: Number of Organs With Metastasis by Tumour EGFR Mutation Status
Description: Summary of number of organs with metastasis. Only participants with at least 1 organ with metastasis are included.
Time Frame: At Screening
Population: Tumour Evaluable Population
Measure: Mean (Standard Deviation); unit: Number
Arm/Group | EGFR Mutation Positive | EGFR Mutation Negative
Number analyzed (Participants) | 925 | 1537
Number | 1.8 (1.05) | 1.6 (0.91)

19. Secondary Outcome: Demographics and Disease Characteristics by Plasma EGFR Mutation Status
Description: as for outcome 16
Time Frame: At Screening
Population: Plasma Evaluable Population
Measure: Number; unit: Participants
Arm/Group | EGFR Mutation Positive | EGFR Mutation Negative
Number analyzed (Participants) | 462 | 2232
Participants
  Histology: Adenocarcinoma | 397 | 1417
  Histology: Non-adenocarcinoma | 60 | 794
  Smoking Status: Never-Smoker | 298 | 835
  Smoking Status: Ever-Smoker | 164 | 1397
  Gender: Male | 228 | 1575
  Gender: Female | 234 | 657
  Region: Asia Pacific | 375 | 1378
  Region: Russia | 87 | 854
  Age: <=65 | 337 | 1454
  Age: >65 | 125 | 778
  WHO Performance Status: 0-1 | 400 | 1956
  WHO Performance Status: 2 | 43 | 237
  Current Disease Status: IIIA | 23 | 257
  Current Disease Status: IIIB | 32 | 378
  Current Disease Status: IV | 407 | 1597
  Number of Organs with Metastasis = 1 | 167 | 956
  Number of Organs with Metastasis = 2 | 120 | 420
  Number of Organs with Metastasis = 3 | 67 | 155
  Number of Organs with Metastasis = 4 | 37 | 57
  Number of Organs with Metastasis = 5 | 12 | 17
  Number of Organs with Metastasis = 6 | 2 | 2
  Number of Organs with Metastasis = 7 | 3 | 0
Statistical Analysis 1: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0009, Regression Stepwise — Age: <=65 vs. >65; 10% Significance Level for entry criteria; Wald Chi Square Statistic = 11.1060
Statistical Analysis 2: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0009, Regression Stepwise — Age: <=65 vs. >65; 10% Significance Level for model entry; Odds Ratio (OR) = 1.561
Statistical Analysis 3: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0001, Regression Stepwise — Number of Organs with Metastisis; 10% Significance Level for entry criteria; Wald Chi Square Statistic = 34.1075
Statistical Analysis 4: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0001, Regression Stepwise — Number of Organs with Metastisis; 10% significance level for model entry; Odds Ratio (OR) = 1.386
Statistical Analysis 5: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0002, Regression Stepwise — Histology: Adenocarcinoma vs. Non-adenocarcinoma; 10% Significance Level for entry criteria; Wald Chi Square Statistic = 14.0806
Statistical Analysis 6: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0002, Regression Stepwise — Histology: Adenocarcinoma vs. Non-adenocarcinoma; 10% Significance Level for model entry; Odds Ratio (OR) = 1.955
Statistical Analysis 7: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0001, Regression Stepwise — Smoking Status: Never-smoker vs. Ever-smoker; 10% Significance Level for entry criteria; Wald Chi Square Statistic = 33.8574
Statistical Analysis 8: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0001, Regression Stepwise — Smoking Status: Never-smoker vs. Ever-smoker; 10% Significance Level for model entry; Odds Ratio (OR) = 2.077
Statistical Analysis 9: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0001, Regression Stepwise — Region: Asia Pacific vs. Russia; 10% Significance Level for entry criteria; Wald Chi Square Statistic = 21.2537
Statistical Analysis 10: Comparison: EGFR Mutation Positive vs EGFR Mutation Negative; Test type: Superiority or Other; p = 0.0001, Regression Stepwise — Region: Asia Pacific vs. Russia; 10% Significance Level for model entry; Odds Ratio (OR) = 2.084

20. Secondary Outcome: Time Since First NSCLC Diagnosis by Plasma EGFR Mutation
Description: Number of months since the first diagnosis of NSCLC from informed consent date.
Time Frame: At Screening
Population: Plasma Evaluable Population
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | EGFR Mutation Positive | EGFR Mutation Negative
Number analyzed (Participants) | 462 | 2232
Months | 2.2 (7.99) | 3.0 (11.09)

21. Secondary Outcome: Number of Organs With Metastasis by Plasma EGFR Mutation Status
Description: Summary of number of organs with metastasis. Only participants with at least 1 organ with metastasis are included.
Time Frame: At Screening
Population: Plasma Evaluable Population
Measure: Mean (Standard Deviation); unit: Number
Arm/Group | EGFR Mutation Positive | EGFR Mutation Negative
Number analyzed (Participants) | 408 | 1607
Number | 2.1 (1.21) | 1.6 (0.89)

22. Secondary Outcome: First Line Treatment Choice by Asia Pacific Country
Time Frame: At Screening
Population: Tumour Evaluable Population
Measure: Number; unit: Participants
Arm/Group | China | Taiwan | South Korea | Australia | Thailand | Singapore | Malaysia | Indonesia | Russia
Number analyzed (Participants) | 1391 | 271 | 62 | 58 | 87 | 100 | 49 | 273 | 924
Participants
  Systemic Anticancer Treatment: Yes | 1151 | 218 | 44 | 45 | 65 | 87 | 29 | 174 | 641
  Systemic Anticancer Treatment: No | 240 | 53 | 18 | 13 | 22 | 13 | 20 | 99 | 283
  Afatinib | 0 | 4 | 1 | 3 | 0 | 10 | 0 | 0 | 13
  Bevacizumab | 5 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
  Carboplatin | 273 | 2 | 10 | 26 | 52 | 23 | 10 | 100 | 235
  Cetuximab | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cisplatin | 424 | 11 | 15 | 3 | 7 | 9 | 12 | 0 | 301
  Crizotinib | 7 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
  Docetaxel | 77 | 18 | 0 | 0 | 1 | 0 | 0 | 0 | 19
  Erlotinib | 21 | 46 | 2 | 5 | 0 | 16 | 0 | 0 | 4
  Etoposide | 12 | 0 | 0 | 2 | 3 | 0 | 0 | 11 | 244
  Gefitinib | 137 | 65 | 6 | 3 | 1 | 21 | 4 | 73 | 33
  Gemcitabine | 284 | 14 | 5 | 25 | 9 | 5 | 22 | 1 | 46
  Icotinib | 55 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Paclitaxel | 133 | 12 | 9 | 4 | 46 | 4 | 0 | 18 | 166
  Pemetrexed | 332 | 25 | 9 | 0 | 0 | 25 | 1 | 0 | 28
  Vincristine | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Vinorelbine | 41 | 22 | 0 | 1 | 0 | 1 | 2 | 0 | 4
  Investigational agent | 17 | 0 | 2 | 2 | 0 | 2 | 0 | 0 | 0
  Other Chemotherapy | 142 | 5 | 1 | 1 | 2 | 0 | 0 | 0 | 44
  Surgery: Yes | 8 | 6 | 1 | 0 | 0 | 1 | 1 | 0 | 12
  Surgery: No | 1383 | 265 | 61 | 58 | 87 | 99 | 48 | 273 | 912
  Radiotherapy: Yes | 62 | 26 | 14 | 14 | 3 | 11 | 17 | 7 | 72
  Radiotherapy: No | 1329 | 245 | 48 | 44 | 84 | 89 | 32 | 266 | 852
  Other: Yes | 33 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 8
  Other: No | 1358 | 271 | 62 | 56 | 87 | 100 | 49 | 273 | 916

23. Secondary Outcome: First Line Treatment Choice by Asia Pacific Country by Tumour EGFR Mutation Status
Time Frame: At Screening
Population: Tumour Evaluable Population
Measure: Number; unit: Participants
Groups:
- China-Mutation Status Positive: Subjects in China that meet I/E and population criteria, who had a Positive Mutation Status.
- China-Mutation Status Negative: Subjects in China that meet I/E and population criteria, who had a Negative Mutation Status.
- Taiwan-Mutation Status Positive: Subjects in Taiwan that meet I/E and population criteria, who had a Positive Mutation Status.
- Taiwan-Mutation Status Negative: Subjects in Taiwan that meet I/E and population criteria, who had a Negative Mutation Status.
- South Korea-Mutation Status Positive: Subjects in South Korea that meet I/E and population criteria, who had a Positive Mutation Status.
- South Korea-Mutation Status Negative: Subjects in South Korea that meet I/E and population criteria, who had a Negative Mutation Status.
- Australia-Mutation Status Positive: Subjects in Australia that meet I/E and population criteria, who had a Positive Mutation Status.
- Australia-Mutation Status Negative: Subjects in Australia that meet I/E and population criteria, who had a Negative Mutation Status.
- Thailand-Mutation Status Positive: Subjects in Thailand that meet I/E and population criteria, who had a Positive Mutation Status.
- Thailand-Mutation Status Negative: Subjects in Thailand that meet I/E and population criteria, who had a Negative Mutation Status.
- Singapore-Mutation Status Positive: Subjects in Singapore that meet I/E and population criteria, who had a Positive Mutation Status.
- Singapore-Mutation Status Negative: Subjects in Singapore that meet I/E and population criteria, who had a Negative Mutation Status.
- Malaysia-Mutation Status Positive: Subjects in Malaysia that meet I/E and population criteria, who had a Positive Mutation Status.
- Malaysia-Mutation Status Negative: Subjects in Malaysia that meet I/E and population criteria, who had a Negative Mutation Status.
- Indonesia-Mutation Status Positive: Subjects in Indonesia that meet I/E and population criteria, who had a Positive Mutation Status.
- Indonesia-Mutation Status Negative: Subjects in Indonesia that meet I/E and population criteria, who had a Negative Mutation Status.
- Russia-Mutation Status Positive: Subjects in Russia that meet I/E and population criteria, who had a Positive Mutation Status.
- Russia-Mutation Status Negative: Subjects in Russia that meet I/E and population criteria, who had a Negative Mutation Status.
Arm/Group | China-Mutation Status Positive | China-Mutation Status Negative | Taiwan-Mutation Status Positive | Taiwan-Mutation Status Negative | South Korea-Mutation Status Positive | South Korea-Mutation Status Negative | Australia-Mutation Status Positive | Australia-Mutation Status Negative | Thailand-Mutation Status Positive | Thailand-Mutation Status Negative | Singapore-Mutation Status Positive | Singapore-Mutation Status Negative | Malaysia-Mutation Status Positive | Malaysia-Mutation Status Negative | Indonesia-Mutation Status Positive | Indonesia-Mutation Status Negative | Russia-Mutation Status Positive | Russia-Mutation Status Negative
Number analyzed (Participants) | 567 | 824 | 130 | 141 | 14 | 48 | 17 | 41 | 25 | 62 | 55 | 45 | 17 | 32 | 116 | 157 | 110 | 814
Participants
  Systemic Anticancer Treatment? Yes | 499 | 652 | 122 | 96 | 12 | 32 | 13 | 32 | 19 | 46 | 54 | 33 | 10 | 19 | 80 | 94 | 86 | 555
  Systemic Anticancer Treatment? No | 68 | 172 | 8 | 45 | 2 | 16 | 4 | 9 | 6 | 16 | 1 | 12 | 7 | 13 | 36 | 63 | 24 | 259
  Afatinib | 0 | 0 | 4 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 0 | 0 | 13 | 0
  Bevacizumab | 1 | 4 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Carboplatin | 96 | 177 | 0 | 2 | 1 | 9 | 1 | 25 | 16 | 36 | 5 | 18 | 3 | 7 | 8 | 94 | 28 | 207
  Cisplatin | 123 | 301 | 2 | 9 | 0 | 15 | 0 | 3 | 2 | 5 | 1 | 8 | 3 | 9 | 0 | 0 | 15 | 286
  Crizotinib | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3
  Docetaxel | 19 | 58 | 3 | 15 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 16
  Erlotinib | 17 | 4 | 43 | 3 | 2 | 0 | 5 | 0 | 0 | 0 | 16 | 0 | 0 | 0 | 0 | 0 | 3 | 1
  Etoposide | 1 | 11 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 3 | 8 | 18 | 226
  Gefitinib | 127 | 10 | 65 | 0 | 6 | 0 | 3 | 0 | 0 | 1 | 21 | 0 | 4 | 0 | 73 | 0 | 24 | 9
  Gemcitabine | 61 | 223 | 1 | 13 | 0 | 5 | 1 | 24 | 3 | 6 | 1 | 4 | 6 | 16 | 1 | 0 | 2 | 44
  Icotinib | 50 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Paclitaxel | 37 | 96 | 2 | 10 | 0 | 9 | 0 | 4 | 13 | 33 | 2 | 2 | 0 | 0 | 4 | 14 | 18 | 148
  Pemetrexed | 139 | 193 | 0 | 25 | 1 | 8 | 0 | 0 | 0 | 0 | 3 | 22 | 0 | 1 | 0 | 0 | 1 | 27
  Vincristine | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Vinorelbine | 14 | 27 | 3 | 19 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 4
  Investigational Agent | 15 | 2 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Other Chemotherapy | 52 | 90 | 1 | 4 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 41
  Cetuximab | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Surgery: Yes | 2 | 6 | 5 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 10
  Surgery: No | 565 | 818 | 125 | 140 | 14 | 47 | 17 | 41 | 25 | 62 | 55 | 44 | 17 | 31 | 116 | 157 | 108 | 804
  Radiotherapy: Yes | 21 | 41 | 2 | 24 | 3 | 11 | 3 | 11 | 2 | 1 | 6 | 5 | 6 | 11 | 2 | 5 | 7 | 65
  Radiotherapy: No | 546 | 783 | 128 | 117 | 11 | 37 | 14 | 30 | 23 | 61 | 49 | 40 | 11 | 21 | 114 | 152 | 103 | 749
  Other: Yes | 14 | 19 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7
  Other: No | 553 | 805 | 130 | 141 | 14 | 48 | 15 | 41 | 25 | 62 | 55 | 45 | 17 | 32 | 16 | 157 | 109 | 807

ADVERSE EVENTS:
Description: Not applicable - no safety data collected in the study
Arm/Group | China | Taiwan | South Korea | Australia | Thailand | Singapore | Malaysia | Indonesia | Russia
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days